CLINICAL TRIAL: NCT03540693
Title: Fat Taste Sensory Study
Acronym: FaTSS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Illinois at Urbana-Champaign (Other)
Collaborators: Carle Foundation Hospital (Other)
Responsible Party: Principal Investigator, Marta Yanina Pepino de Gruev, Assisstant Professor of Ingestive Behavior, University of Illinois at Urbana-Champaign
Other Study IDs: 18439
Record Dates: First submitted 2018-05-04; First posted 2018-05-30 (Actual); Last update posted 2021-04-28 (Actual); Status verified 2021-04

CONDITIONS: Bariatric Surgery Candidate; Bariatric Surgical Procedure
Keywords: Bariatric surgery; gastric bypass surgery; sleeve gastrectomy; laparoscopic gastric banding; food preferences; flavor perception
MeSH Terms: conditions — Food Preferences

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples With DNA — DNA extracted from saliva
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- RYGB-longitudinal: Longitudinal group of subjects studied before and after Roux-n-Y gastric bypass surgery
  Interventions: Procedure: RYGB
- SG_longitudinal: Longitudinal group of subjects studied before and after sleeve gastrectomy surgery
  Interventions: Procedure: SG
- LAGB_longitudinal: Longitudinal group of subjects studied before and after laparoscopic gastric banding surgery
  Interventions: Procedure: LAGB
- Weight-loss success: Subjects who lost ≥40% body weight by 2-5 years post-surgery
  Interventions: Procedure: RYGB; Procedure: SG
- Weight-loss failure: Subjects who lost <25% body weight (or lost more but then regain weight so that now are at <25%) by 2-5 years post-surgery
  Interventions: Procedure: RYGB; Procedure: SG

INTERVENTIONS:
Procedure: RYGB — RYGB-weight loss surgery
  Groups: RYGB-longitudinal; Weight-loss failure; Weight-loss success
Procedure: SG — SG- weight loss surgery
  Groups: SG_longitudinal; Weight-loss failure; Weight-loss success
Procedure: LAGB — LAGB- weight loss surgery
  Groups: LAGB_longitudinal

SUMMARY:
Fat is the most energy dense macronutrient and consuming fat has been positively correlated to obesity. Individuals afflicted with obesity crave fat more frequently, have a higher preference for fatty taste, and consume a higher quantity of fatty foods. People who have undergone Roux-en-Y Gastric Bypass (RYGB) or Sleeve Gastrectomy (SG) weight-loss surgeries dramatically decrease their fat preferences and consumption of fat, at least within the first year after surgery. These surgeries are very effective in helping people lose weight over the first couple of years; however, approximately 30% of those who undergo these surgeries start regaining weight after the second year mark. Why some people are able to keep the weight off long-term but others are unable to is unclear. In addition, it is well-known that fat can modify the flavor of foods and flavor plays a critical role in consumption, as well as in responses that gear up the body to consume the food. These are known as cephalic phase responses and include neural, physiological, and hormonal aspects. The main goals of the study are twofold: 1) To test the immediate effects of RYGB surgery, SG surgery, and laparoscopic gastric banding (LAGB) surgery (a weight loss control group) on fat preferences and sensory perception, and 2) to compare fat preferences and sensory perception between those who are able to achieve sustained weight loss 2-5 years after RYGB or SG surgery and those who either regained weight or did not lose the desired amount.

DETAILED DESCRIPTION:
For the first goal, the investigators will assess a longitudinal group of subjects both before RYGB surgery (n=15) SG surgery (n=15), and LAGB surgery (n=15), and then again after they lose ~16% of their body weight post-surgery in the fed and the fasted state. the investigators will also study the same variables in a cross-sectional design consisting of two groups: a weight success group (n=30) and a weight failure group (n=30) 2-5 years post RYGB or SG surgery. The weight success group will include subjects who lost ≥40% body weight by 2-5 years post-surgery and the weight failure group will include subjects who lost <25% body weight by 2-5 years post-surgery. In addition, the investigators will also explore the extent to which fat preferences and sensory perception in these subjects are affected by flavor related genes.

ELIGIBILITY:
Inclusion Criteria:

* Women and men, 18-64 years of age, all races
* Subjects must be scheduled to undergo Roux-en-Y Gastric Bypass surgery (RYGB), Sleeve Gastrectomy surgery (SG), or laparoscopic gastric banding surgery (LAGB) and be available to be tested both pre- and post-surgery or must have undergone RYGB or SG surgery between 2-5 (i.e. at least two years ago and not more than 5) years ago and have a current weight loss that is ≥40% of body weight pre-surgery or <25% of body weight pre-surgery.

Exclusion Criteria:

* Smoking tobacco related cigarettes or having quit smoking less than 6 months ago
* Pregnant or breastfeeding
* Are experiencing significant organ dysfunction
* Take medications that could influence research results
* Have any psychiatric illness or disorder that could influence compliance or completion of the study
* History of chronic rhinitis
* Had a diagnosis of or are taking medicine to treat diabetes
* Inflammatory intestinal disease
* Subjects who underwent RYGB or SG between 2-3 years ago and have a current weight loss that is <40% and ≥25% of their body weight pre-surgery.
* Subjects must find the taste of the food to be sham-fed acceptable (e.g. cream cheese, etc.).

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: 1) Participants scheduled to undergo Roux-en- Y Gastric Bypass (RYGB) surgery, Sleeve Gastrectomy (SG) surgery, or Laparoscopic Gastric Banding (LAGB) surgery or 2) have had RYGB or SG surgery 2-5 years ago and fall into one of two groups: Group 2a) as a result of the surgery she/he lost ≥40% of pre-surgery body weight and was able to keep it off until now or Group 2b) lost <25% of pre-surgery body weight or lost more but regained the weight.
Sampling Method: Non-Probability Sample
Enrollment: 105 (Estimated)
Dates: Start 2018-04-06 (Actual); Primary Completion 2023-04-06 (Estimated); Study Completion 2023-07-06 (Estimated)

PRIMARY OUTCOMES:
Flavor perception | 3-6 months
  Changes in perception of flavor intensity in the general label magnitude scale (in mm)
Flavor preference | 3-6 months
  Changes in perception of hedonic value in the hedonic version of the general label magnitude scale (in mm)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Illinois at Urbana Champaign, Urbana, Illinois, United States

IPD SHARING:
Plan to Share IPD: No